CLINICAL TRIAL: NCT03553680
Title: An Emotion-Focused Psychosocial Intervention for Improved Glycemic Control in T2D Patients: A Pilot Study
Brief Title: An Emotion-Focused Intervention for Glycemic Control in T2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0635
Record Dates: First submitted 2018-05-16; First posted 2018-06-12 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2018-05

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: Emotion-Focused CBT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion-Focused CBT (Experimental): Ten CBT sessions with a therapist.
  Interventions: Behavioral: Emotion-Focused CBT
- Wait List (No Intervention): Three visits for assessments only over the same time period of the Experimental Arm.

INTERVENTIONS:
Behavioral: Emotion-Focused CBT — 10 CBT Sessions to improve emotional regulation and emotional intelligence.
  Arms: Emotion-Focused CBT

SUMMARY:
The primary aim of this proposed project is to collect pilot data using an Emotion-Focused CBT Psycho-social Intervention i individuals with T2D to obtain the effect sizes on hypothesized changes in Negative Emotionality, Diabetes Distress, and HbA1c values that will be needed for a more appropriately sized clinical trial for an RO1 submission to the National Institutes of Health.

DETAILED DESCRIPTION:
Our interest in aberrant Emotional Regulation / Emotional Intelligence in Type 2 Diabetes stems from observations that while many patients with Type 2 Diabetes have greater incidence of mood and anxiety (and even anger) disorders than controls, targeting psychiatric conditions, such as depression, is not sufficient to improve glycemic control in patients with diabetes. Thus, the key issue for such patients is not what specific psychiatric disorder they have, but the presence of an impairment in the fundamental regulation of emotional regulation and in how such individuals modulate their emotional response to aversive events in their lives (e.g., emotional intelligence), now suggested by a recent study. As part of a new study, we examined the relationship between glycemic control (HbA1c) and Emotional Experience (ER-Exp) and Skill at Emotional Regulation (ER-Skill) in 100 adult patients with Type 2 Diabetes. We found significant relationships between ER-Exp and ER-Skill and HbA1c levels that accounted for nearly 24% of the variance in HbA1c levels. These relationships with HbA1c levels remained even after accounting for other relevant behavioral variables such as depression/anxiety scores and diabetes self-care/literacy scores. Accordingly, the tendency of an individual to have intense emotional responses (higher scores on ER-Exp), and/or to have a reduced ability to understand/modulate one's emotions in order to cope with daily stresses/threats (lower scores on ER-Skill), may well be linked with poor glycemic control (HbA1c) in adult patients with Type 2 Diabetes. If so, it will be important to develop psycho-social methods to improve ER-Exp and DR-Skill in Type 2 Diabetes patients to determine if one can improve aberrant Emotional Regulation (ER-Exp/ER-Skill), Diabetes Distress (DD), and HbA1c (A1c) levels as suggested by treatment studies showing that such treatment can improve ER-Skill with a sustained reduction in A1c levels in Type 2 Diabetes for up to nine months. Supporting these findings are data from a recent study showing that increasing positive emotion reduces (and increasing negative emotion increases) blood glucose levels, especially in those with poor emotion regulation skills.

Specific Study Objectives:

* Develop an integrated Emotion - Focused Psycho-social EF-CBT) from three (3) existing sources that contain elements to improve ER-Exp and ER-Skill.
* Conduct a pilot study in 10 patients with Type 2 Diabetes with aberrant ER-ER-Exp/ER-Skill and compare treatment outcomes in emotionality, diabetes distress, and in A1c levels with 10 patients with Type 2 Diabetes undergoing treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

1. Receiving care for T2D at Kovler Diabetes Center, at UCM, or in the community.
2. Documented diagnosis of T2D for at least one year.
3. Age: 21-65 years of age.
4. HbA1c > 7.0 (with hemoglobin in the normal range).
5. ER-Exp Screen score of > 29 and/or ER-Skill Screen score < 44.
6. Stable medical co-morbid conditions.
7. Able to read English.
8. Able to give informed consent.

Exclusion Criteria:

1. Documented diagnosis of T2D less than one year.
2. Age: < 21 or > 65 years of age.
3. HbA1c < 7.0 .
4. ER-Exp screen score of < 29 and ER-Skill score =/> 44.
5. Unstable medical co-morbid conditions.
6. Active psychosis or suicidal/homicidal ideation.
7. Not able to read English.
8. Not able to give informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Change in the ER-Exp Score | Baseline, mid-point, and end-point (about 10-12 weeks).
  ER-Exp: Intensity and lability of negative emotion, higher scores indicate greater native emotionality
Change Score in ER-Skill Score | Baseline, ,mid-point and end-point (about 10-12 weeks)
  Skill at emotional regulation (Clarity and Repair). Lower scores indicate reduced skill at modulating negative emotions
Change in HbA1c level | Baseline, mid-point, and end-point (about 10-12 weeks)
  HbA1c levels
Change in Diabetes Distress | Baseline, mid-point, and end-point (about 10-12 weeks)
  Distress at living with and coping with diabetes

SECONDARY OUTCOMES:
Change in Diabetes Self-Care | Baseline, mid-point, and end-point (about 10-12 weeks)
  Self-Care Inventory-Revised: higher scores mean great efforts at self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Emil F Coccaro, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No